CLINICAL TRIAL: NCT01364571
Title: A Phase 1/2 Placebo-controlled, Randomized, Double-blind Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of 3 Ascending Dose Levels Of A 4-antigen Staphylococcus Aureus Vaccine (sa4ag) In Healthy Adults Aged 18 To <65 Years
Brief Title: Evaluation of a Single Vaccination With One of Three Ascending Dose Levels of a 4-Antigen Staphylococcus Aureus Vaccine (SA4Ag) in Healthy Adults Aged 18 to <65 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B3451001; 6123K1-1005 (Other: Alias Study Number)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Staphylococcal Infections
Keywords: Staphylococcus aureus; vaccine; staphylococcal infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): SA4Ag vaccine low dose
  Interventions: Biological: SA4Ag vaccine low dose; Procedure: Blood draw; Procedure: Colonization swab sample
- 2 (Experimental): SA4Ag vaccine mid dose
  Interventions: Biological: SA4Ag vaccine mid dose; Procedure: Blood sample; Procedure: Colonization swab sample
- 3 (Experimental): SA4Ag vaccine high dose
  Interventions: Biological: SA4Ag vaccine high dose; Procedure: Blood draw; Procedure: Colonization swab sample
- 4 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo; Procedure: Blood draw; Procedure: Colonization swab sample

INTERVENTIONS:
Biological: SA4Ag vaccine low dose — Subjects receive 1 intramuscular injection (0.5 mL) of the low dose level of the SA4Ag vaccine.
  Arms: 1
Procedure: Blood draw — Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 1
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various time points throughout the study.
  Arms: 1
Biological: SA4Ag vaccine mid dose — Subjects receive 1 intramuscular injection (0.5 mL) of the mid dose level of the SA4Ag vaccine.
  Arms: 2
Procedure: Blood sample — Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 2
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various time points throughout the study.
  Arms: 2
Biological: SA4Ag vaccine high dose — Subjects receive 1 intramuscular injection (0.5 mL) of the high dose level of the SA4Ag vaccine.
  Arms: 3
Procedure: Blood draw — Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 3
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various time points throughout the study.
  Arms: 3
Biological: Placebo — Subjects receive one intramuscular injection (0.5 mL) of commercially available normal saline.
  Arms: 4
Procedure: Blood draw — Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 4
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various time points throughout the study.
  Arms: 4

SUMMARY:
This is a first-in-human (Phase 1) and Phase 2 study of a single vaccination with one of three dose levels of an investigational vaccine against Staphylococcus aureus (SA4Ag). The main goal of the study is to determine how safe and well tolerated the vaccine is as well as to describe the immune response elicited by the vaccine in healthy adults aged 18 to <65 years. In addition, the study aims to assess the effect of the SA4Ag vaccine on the presence of the Staphylococcus aureus on the skin and within the nose, throat and perineum of healthy adults aged 18 to <65 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to <65 years at enrollment, as determined by medical history, physical examination, and the clinical judgment of the investigator to be eligible for the study. Subjects with preexisting chronic medical conditions determined to be stable may be included.
* Availability for the entire duration of the study, and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including completion of the electronic diary (e-diary) from Day 1 to Day 14 following vaccination(s).
* Ability to be contacted by telephone during study participation.
* All male and female subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control for the duration of the study.

Exclusion Criteria:

* Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization within 3 months before receipt of study vaccine.
* Serious chronic medical disorders and any other disorder that in the investigator's opinion precludes the subject from participating in the study
* Donation of blood volume of 250 mL or greater (excluding protocol-required blood collection), or donation of plasma within 3 months prior to enrollment.
* Bleeding condition associated with prolonged bleeding time that may contraindicate intramuscular injection or blood draw including subjects taking anticoagulant, antiplatelet and/or antithrombotic agents except for low-dose daily aspirin within 30 days before enrollment through 1 month post-vaccination.
* Any contraindication to vaccination or vaccine components.
* Immunocompromised persons and subjects currently on immunosuppressive therapy or with a history of immunosuppressive therapy, including chemotherapy agents or long term systemic corticosteroids.
* Previous administration of S. aureus vaccination.
* Any infection proven or suspected to be caused by S. aureus within 6 months preceding study vaccination.
* Receipt of blood products or immunoglobulins (including monoclonal antibodies) within 12 months before enrollment through conclusion of the study.
* Participation in other investigational or interventional studies within 30 days before the current study begins and/or during study participation.
* Subjects who are investigational site staff members or subjects who are immediate family members (1st degree relatives) of investigational site staff members or Pfizer employees directly involved in the conduct of the trial.
* Residence in a nursing home or long-term care facility or requirement for semiskilled nursing care.
* For Phase 1 subjects only, any abnormality in screening hematology, coagulation and/or blood chemistry laboratory values.
* Women who are pregnant (as determined by urine pregnancy test) or breastfeeding.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 456 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects reporting local reactions (size of redness and/or swelling and severity of pain at the injection site) and severity of the local reactions as self-reported on electronic diaries (e-diaries) | 14 days
Number and proportion of subjects reporting solicited systemic events (fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, new or worsening joint pain) and severity of solicited systemic events self-reported on electronic diaries | 14 days
Number and proportion of subjects reporting unsolicited AEs and serious adverse events (SAEs) categorized according to the Medical Dictionary for Regulatory Activities (MedDRA) | 1 month (AEs), 6 months (SAEs)
Number and proportion of Phase 1 subjects with abnormal hematology, coagulation and blood chemistry lab assessments; number and proportion of Phase 1 subjects with grading shifts in hematology, coagulation and blood chemistry laboratory assessments. | 14 days
Proportion of subjects achieving antibody responses to specific antigens with results greater than or equal to thresholds specific to each of the 4 antigens in the vaccine based on immunoglobulin-binding and/or opsonophagocytic activity assays. | 1 month

SECONDARY OUTCOMES:
Immunoglobulin concentrations for each antigen at each applicable blood sampling time point, | various, up to 12 months
Opsonophagocytic activity (OPA) titers at each applicable blood sampling time point, | 1 month
Immunoglobulin geometric mean fold rise (GMFR) for each antigen | 1 month
Geometric mean fold rise on opsonophagocytic activity assay titers | 1 month
Proportion of subjects achieving antibody responses to specific antigens with results greater than or equal to thresholds specific to each of the 4 antigens in the vaccine at at each applicable visit | various, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- United States (15):
  - Broward Research Group, Hollywood, Florida
  - Miami Research Associates, South Miami, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - SNBL Clinical Pharmacology Center, Inc., Baltimore, Maryland
  - Prism Research, Saint Paul, Minnesota
  - Buffalo Clinical Research Center, LLC, Buffalo, New York
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Roberta Braun, M.D., Austin, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas

REFERENCES:
- [Derived] Creech CB, Frenck RW, Fiquet A, Feldman R, Kankam MK, Pathirana S, Baber J, Radley D, Cooper D, Eiden J, Gruber WC, Jansen KU, Anderson AS, Gurtman A. Persistence of Immune Responses Through 36 Months in Healthy Adults After Vaccination With a Novel Staphylococcus aureus 4-Antigen Vaccine (SA4Ag). Open Forum Infect Dis. 2019 Dec 24;7(1):ofz532. doi: 10.1093/ofid/ofz532. eCollection 2020 Jan. PMID 31993453
- [Derived] Frenck RW Jr, Creech CB, Sheldon EA, Seiden DJ, Kankam MK, Baber J, Zito E, Hubler R, Eiden J, Severs JM, Sebastian S, Nanra J, Jansen KU, Gruber WC, Anderson AS, Girgenti D. Safety, tolerability, and immunogenicity of a 4-antigen Staphylococcus aureus vaccine (SA4Ag): Results from a first-in-human randomised, placebo-controlled phase 1/2 study. Vaccine. 2017 Jan 5;35(2):375-384. doi: 10.1016/j.vaccine.2016.11.010. Epub 2016 Dec 1. PMID 27916408